CLINICAL TRIAL: NCT06854185
Title: Feasibility of the "Paso a Paso" Weight Loss Program for Mexican & Central American Patients With Metabolic Dysfunction Associated Steatotic Liver Disease(MASLD)
Brief Title: Feasibility of the Paso Program for Patients With Metabolic Dysfunction Associated Steatotic Liver Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Maya Balakrishnan, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-55723; K23MD016955 (NIH)
Record Dates: First submitted 2025-02-21; First posted 2025-03-03 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Dysfunction Associated Steatotic Liver Disease; Overweight (BMI > 25); Metabolic Syndrome
Keywords: metabolic dysfunction associated steatotic liver disease; adapted weight loss intervention; weight loss; intervention feasibility; behavior change; metabolic syndrome; overweight/obesity
MeSH Terms: conditions — Overweight; Metabolic Syndrome; Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: This is a single arm trial testing the feasibility of the behavioral weight loss program. All study participants will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): All participants will receive the intervention, which is a behavioral weight loss program called "Paso a Paso: Rumbo a Un Higado Sano" ("Paso Program").
  Interventions: Behavioral: Paso Program

INTERVENTIONS:
Behavioral: Paso Program — The Paso Program is a behavioral weight loss program. It consists of a series of 16 one-hour-long semi-structured group counseling sessions led by a health educator every 1-2 weeks over 26 weeks. Each session has a curriculum with a counselor's guide and patient facing materials, covers specific topics (eating, physical activity, behavioral change strategies). Teaching methods include discussions, practice activities, demonstrations. The program is delivered to groups of 8 to 14 participants, classes are offered primarily in-person with the option of virtual attendance.
  Other Names: Paso a Paso: Rumbo a Un Higado Sano; Step by Step: Journey to a Healthy Liver

SUMMARY:
The purpose of this study is to learn whether the Paso weight loss program is feasible for Mexican and Central American patients with fatty liver disease. In addition, the investigators will also look at whether the program improves weight loss, fatty liver disease, physical activity, diet, and family support among patients.

DETAILED DESCRIPTION:
Weight loss is an important part of treating fatty liver disease. The investigators have developed a weight loss program for Mexican and Central American patients with fatty liver disease (also known as Metabolic Dysfunction Associated Steatotic Liver Disease). The name of the weight loss program is "Paso a Paso: Rumbo a Un Higado Sano" / "Step by Step: Journey to a Healthy Liver."

The purpose of this study is to learn whether the Paso weight loss program is acceptable to patients and feasible to participate in.

Participants who join the study will participate in a 6 month weight loss program, consisting of 16 1-hour group counseling classes that teach about healthy eating, physical activity, and behavioral strategies to break old habits and create new ones. Participants are required to attend 4 classes in person, and the remainder can be attended in person or virtually.

The program classes are offered at 5 locations across Houston. Participants can choose the location most convenient, and are then assigned to that location, along with other participants who also choose that location, for the duration of the program.

Study participants will be asked to complete questionnaires and testing for the study at 4 time points over 1 year: before starting the program, in the middle of the program, at the end of the program, and 6 months after the program ends. All questionnaires and testing are done during regular clinic visits, during program sessions, or over the phone. The testing includes questionnaires, measurement of your weight and muscle strength, and an optional fibroscan (ultrasound) of the liver. In addition, data about medical history and blood testing will be recorded from participants' medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with MASLD (defined per guideline based diagnostic criteria: evidence of steatosis with at least 1 metabolic syndrome feature)
2. Self-reported Mexican or Central American ethnicity
3. Age between 18 and 70 years
4. BMI≥25kg/m2
5. Able to read and write English and/or Spanish

Exclusion Criteria:

1. ≥5% weight loss over the prior 3 months
2. HbA1c ≥9.0% within 30 days of weight loss program initiation*
3. History of bariatric surgery
4. Advanced liver disease, defined as:

   platelet count < 150,000, serum albumin <3.5 g/dL, except as explained by non-hepatic causes. INR >1.4 unless due to therapeutic anticoagulants or laboratory error. Total bilirubin ≥2 mg/dL (unless explained by Gilbert Syndrome). Presence of esophageal varices,
5. Any history of liver disease decompensations** or hepatocellular carcinoma,
6. History of any organ transplant (including liver transplant)
7. Active HCV infection (defined as HCV Ab positive with detectable viral load)*, Hepatitis B infection (defined as positive HBsAg) and/or other etiologies of chronic liver disease (AIH, PBC, Wilson disease, PSC) or acute hepatic injury.
8. Ongoing heavy alcohol use defined as 320-420grams/week
9. SGLT2 inhibitor or Glucagon-like peptide 1 (GLP-1) agonist therapy for diabetes treatment (e.g., exenatide, liraglutide, lixisenatide, albiglutide, dulaglutide, semaglutide, and albiglutide) or for weight loss (e.g., semaglutide at doses up to 2.4 mg subcutaneous weekly) must be at a stable dose for at least 6 months prior to study entry with stable weight (defined as <5% weight loss in the 12 weeks prior to study entry)*
10. Pioglitazone is allowed if on a stable dose for 3 months prior to study entry
11. current pregnancy/nursing or planned pregnancy
12. conditions limiting dietary calorie reduction or physical activity
13. Active cancer, except for example non-melanoma skin cancers or cancers that have clearly been cured, stable and being monitored by primary doctor or oncologist without active treatment, or carries an excellent prognosis (e.g., Stage 1 cervical cancer)
14. unstable cardiac disease
15. intestinal resection or malabsorption disorders
16. life expectancy<2 years
17. competing serious medical or psychiatric comorbidity
18. HIV infection
19. History of noncompliance (>3 primary care, endocrine, and/or hepatology clinic no-shows in the past year)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasbility | 6 months
  Average attendance > 8 sessions across participants

SECONDARY OUTCOMES:
change in percent weight | baseline to 6 months
  average percent change in weight
change in absolute weight | baseline to 6 months
  Average absolute weight change (kg)
change in muscle strength | baseline to 6 months
  Average change, measured by hand grip dynamometry
change in liver stiffness | baseline to 6 months
  Average Change in liver stiffness values assessed by transient elastography
change in liver CAP | baseline to 6 months
  Average change in continued attenuation parameter assessed by transient elastography
change in liver enzymes | baseline to 6 months
  Average change in transaminases
change in hemoglobin A1C | baseline to 6 months
  Average change in hemoglobin a1c
change in diet quality | baseline to 6 months
  Average change in Healthy Eating Index assessed by diet history questionnaire III. The Healthy eating score ranges from 0 to 100. A higher number means a healthier diet quality.
change in daily calorie intake | baseline to 6 months
  change in average daily calorie intake assessed by DHQIII
change in fat intake | baseline to 6 months
  Change in average fat intake assessed by DHQIII
change in alcohol intake | baseline to 6 months
  Change in alcohol intake, assessed by AUDIT-C
change in average weekly minutes of moderate-to-vigorous physical activity | baseline to 6 months
  Change in average time spent doing moderate to vigorous physical activity every week assessed by actigraphy
change in average daily steps | baseline to 6 months
  change in average daily steps assessed by actigraphy
change in quality of life | baseline to 6 months
  change in quality of life assessed by a questionnaire called "Patient-Reported Outcomes Measurement Information System - Global score"
Change in perception of metabolic dysfunction associated steatotic liver disease | baseline to 6 months
  Change in average composite score, Illness perception questionnaire
Change in perceived treatment efficacy | baseline to 6 months
  Change in average composite score, treatment efficacy questionnaire
Change in dietary self-efficacy | baseline to 6 months
  Change in dietary self-efficacy assessed using Schwarzer & Renner scale
Change in physical activity self-efficacy | baseline to 6 months
  Change in physical activity self-efficacy assessed using Schwarzer & Renner scale
Change in social support for diet | baseline to 6 months
  Change in diet social support assessed using Sallis perceived social support scale
Change in social support for physical activity | baseline to 6 months
  Change in physical activity social support assessed using Sallis perceived social support scale
Change in perceived stress | baseline to 6 months
  assessed by perceived stress scale
change in % weight | baseline to 1 year
  average % change in weight
change in absolute weight | baseline to 1 year
  Average absolute weight change (kg)
change in muscle strength | baseline to 1 year
  Average change, measured by hand grip dynamometry
change in liver stiffness and CAP | baseline to 1 year
  Average change in liver stiffness and continued attenuation parameter assessed by transient elastography
change in liver enzymes | baseline to 1 year
  Average change in transaminases
change in lipids | baseline to 1 year
  Average change in lipids
change in physical activity level | baseline to 1 year
  Change in physical activity category assessed by the International Physical Activity Questionnaire. This questionnaire estimates the estimated resting energy expenditure and can categorize people's physical activity level as low, moderate, or high.
change in physical activity level | baseline to 6months
  Change in physical activity category assessed by the International Physical Activity Questionnaire. This questionnaire estimates the estimated resting energy expenditure and can categorize people's physical activity level as low, moderate, or high.
Change in dietary self-efficacy | baseline to 1 year
  Change in dietary self-efficacy assessed using Schwarzer & Renner scale
Change in physical activity self-efficacy | baseline to 1 year
  Change in physical activity self-efficacy assessed using Schwarzer & Renner scale
Change in social support for diet | baseline to 1 year
  Change in diet social support assessed using Sallis perceived social support scale
Change in social support for physical activity | baseline to 1 year
  Change in physical activity social support assessed using Sallis perceived social support scale
change in average weekly minutes of moderate-to-vigorous physical activity | baseline to 1 year
  Change in average time spent doing moderate to vigorous physical activity every week assessed by actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Maya Balakrishnan, Principal Investigator — Baylor College of Medicine
Locations (1):
- Harris Health - Smith, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This study's primary purpose is to test the feasibility of the Paso program in this pilot single arm study. Therefore, IPD sharing is not planned at this time.

REFERENCES:
- See also: This website provide a description of the Paso program. It also gives study participants electronic access to session materials and meal plans. — https://www.bcm.edu/paso-a-paso-higado-sano

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: IRB protocol report (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT06854185/Prot_SAP_000.pdf
  • Study Protocol: Full protocol (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT06854185/Prot_001.pdf
  • Informed Consent Form: English Consent Form (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT06854185/ICF_002.pdf